CLINICAL TRIAL: NCT06924424
Title: Aponermin, Pomalidomide, Dexamethasone for Patients With Relapsed/ Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, MD, Dr, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-372-001
Record Dates: First submitted 2025-04-06; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma, Neoplasms
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apo-Pd for R/R MM (Experimental): Aponermin10mg/kg d1-5 ivgtt Pomalidomide 4mg d1-21 po Dex 20mg d1;d8;d15 po
  Interventions: Drug: Aponermin, pomalidomide, dexamethasone

INTERVENTIONS:
Drug: Aponermin, pomalidomide, dexamethasone — Three drugs combination for R/R MM. Aponermin, 10mg/kg d1-5 Pomalidomide 4mg d1-21 Dexamethasone 20mg d1,d8,d15 Each treatment cycle is 28 days.

SUMMARY:
This study aims to evaluate the efficacy and safety of a three drug combination therapy of aponermin, pomalidomide, and dexamethasone in the treatment of relapsed or refractory multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

1. RRMM patients who have received 1-3 line treatment;
2. Age above 18 years old, male or female not limited;
3. ECOG score ≤ 2;
4. Expected survival period is greater than 3 months;
5. For female patients, (1) they have been menopausal for at least 24 months before the screening visit, or have undergone surgical contraception; (2) Women with fertility must have two negative urine HCG pregnancy tests within 72 hours before starting to take the study drug; For male patients must agree to absolute abstinence or effective barrier contraception throughout the entire study treatment period until 28 days after the last study drug treatment, and have no sperm donation behavior;
6. The patient understands the purpose and steps of this trial, voluntarily participates in this trial, and signs a written informed consent form.

Exclusion Criteria:

1. Allergic or intolerant to the investigational drug or its components;
2. Received any experimental drug treatment within 4 weeks;
3. Simultaneously suffering from other tumors, or having undergone anti-tumor treatment (including major surgery) in the past 4 weeks;
4. Currently, there are poorly controlled heart diseases, such as heart function grade III or IV (NYAH classification),uncontrolled atrial fibrillation, unstable angina, and myocardial infarction within the 12 months prior to enrollment;
5. Suffering from mental illness;
6. Accompanied by severe lung infection, skin and soft tissue infection, or urinary tract infection;
7. There was a serious thrombotic event before treatment;
8. Unable or unwilling to receive prophylactic antithrombotic therapy;
9. Serious, uncontrolled medical disorders or active infections;
10. Researchers determine situations that are not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response | 4 months
  Overall haematological response after 4 cycles of treatments

SECONDARY OUTCOMES:
PFS | 2 years
  Progression free survival, from initiation of Apo-Pd treatment to the occurrence of disease progression or death
Adverse events | 2 years
  To determine safety of aponermin, pomalidomide and dexamethasone for the treatment of relapsed and refractory multiple myeloma

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No